CLINICAL TRIAL: NCT06054477
Title: A Phase I/II, Open-Label, Multi-Center Study of ALE.C04 as a Single Agent and in Combination With Pembrolizumab in Adult Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Study of ALE.C04 in Patients With Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Reprioritization of Trial
Sponsor: Alentis Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALE.C04.01
Record Dates: First submitted 2023-09-07; First posted 2023-09-26 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: Immunotherapy; Anti-Claudin1; ALE.C04; Phase I/II
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1 will consist of i) a dose escalation of ALE.C04 monotherapy evaluating approximately 3 dose levels of ALE.C04, ii) a dose escalation of ALE.C04 and pembrolizumab combination evaluating approximately 2 dose levels of ALE.C04 and iii) a randomized two RDEs evaluating two dose level of ALE.C04 combined with pembrolizumab to establish Recommended Phase 2 Dose (RP2D).
  Phase 2 will consist of a 1:1 randomized 2 arms comparing ALE.C04 (at the RP2D dose determined in the phase 1) combined to pembrolizumab with pembrolizumab alone.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Dose Escalation (Experimental): ALE.C04 single agent: Three planned doses of ALE.C04 and ALE.C04 in combination with pembrolizumab. Once a certain dose level of ALE.C04 is considered safe and well tolerated, the first cohort of patients receiving ALE.C04 at a lower dose level combined with pembrolizumab will be initiated
  Interventions: Drug: ALE.C04; Drug: Pembrolizumab
- Phase 1 Recommended Dose for Expansion (Experimental): Two ALE.C04 dose levels (higher or lower) will be considered for the combination with pembrolizumab
  Interventions: Drug: ALE.C04; Drug: Pembrolizumab
- Phase 2 Randomized Combination part (Active Comparator): ALE.C04 at RP2D combined to pembrolizumab compared to pembrolizumab monotherapy
  Interventions: Drug: ALE.C04; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ALE.C04 — Q3W
Drug: Pembrolizumab — 200mg Q3W
  Other Names: Keytruda

SUMMARY:
The purpose of this study is to evaluate the safety profile of ALE.C04 monotherapy and in combination with pembrolizumab, to characterize pharmacokinetics profile of ALE.C04, recommended Phase II dose (RP2D) for ALE.C04 in combination with pembrolizumab and to assess anti-tumor activity of ALE.C04 in combination with pembrolizumab in patients with Head and Neck Cancer.

DETAILED DESCRIPTION:
The study comprises a phase I and a phase II. The phase I dose escalation part for both ALE.C04 monotherapy and in combination with pembrolizumab and a recommended dose for expansion (RDE) part for ALE.C04 in combination with pembrolizumab. The phase II comprises a 1:1 randomized 2 arms assessing ALE.C04 and pembrolizumab given in combination versus pembrolizumab monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consents
2. Be 18 years of age on day of signing informed consent.
3. Have histologically or cytologically confirmed Recurrent or Metastatic (R/M) Head and Neck Squamous Cell Carcinoma (HNSCC) that is considered incurable by local therapies.
4. Have provided tissue for claudin-1 (CLDN1), programmed death ligand-1 (PD-L1) and biomarker analysis in a central Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
5. Have measurable disease based on RECIST 1.1 as determined by the site.
6. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
7. Have results from testing of human papillomavirus (HPV) status for oropharyngeal cancer

Exclusion Criteria:

1. Has progressive disease (PD) within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC (Phase II randomized combination part only).
2. Has had radiation therapy (or other non-systemic therapy) within 2 weeks prior to randomization or patient has not fully recovered (i.e., ≤Grade 1 or at baseline) from adverse events due to a previously administered treatment. Palliative radiotherapy to a limited field is allowed.
3. Severe immune-related adverse events leading to discontinuation of prior immune-oncology agent only for Phase I dose escalation monotherapy and combination and Phase II monotherapy.
4. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
5. Dermatological conditions requiring active pharmacological treatment including psoriasis, atopic dermatitis, excessively dry skin or recurrent conjunctivitis, scleroderma, vitiligo, or any other active autoimmune dermatological disorder.
6. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the clinical study, interfere with the patient's participation for the full duration of the clinical study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
7. Has received prior therapy with an anti-programmed death (PD)-1, anti-PD-L1 or anti-PD-L2 (Phase II randomized combination part only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLT) | 21 days
  Phase I dose escalation
Incidence and severity of adverse events (AEs), serious adverse events (SAEs) | Up to 30 days after last dose - Approximately 4.5 years
  Descriptive statistics will be used to summarize results
Confirmed Objective Response Rate (ORR) by investigators assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 4.5 year
  Proportion of patients with confirmed Complete Response (CR) or Partial Response (PR) according to RECIST 1.1 for Phase II
Confirmed Progression Free Survival (PFS) by Blinded Independent Central Review (BICR) assessment according to RECIST1.1 | Up to 4.5 year
  Time from start of study treatment to first documentation of objective progressive disease (PD) as per RECIST1.1 or to death due to any causes whichever come first during phase II

SECONDARY OUTCOMES:
Confirmed ORR by investigators assessment according to RECIST1.1 | up to 4.5 year
  Proportion of patients with confirmed CR or PR according to RECIST1.1
Confirmed immune Objective Response Rate (iORR) by investigators assessment according to immune RECIST | up to 4.5 year
  Proportion of patients with confirmed immune CR or immune PR according to immune RECIST
Disease Control Rate (DCR) as per investigator assessment according to RECIST1.1 | up to 4.5 years
  Proportion of patients with CR, PR or Stable Disease (SD) according to RECIST1.1
Immune Disease Control Rate (iDCR) as per investigator assessment according to immune RECIST | up to 4.5 years
  Proportion of patients with immune CR, immune PR or immune SD according to immune RECIST
Duration Of Response (DOR) | up to 4.5 years
  The time from first documentation of objective response to the first documentation of PD per RECIST 1.1 or to death due to any cause, whichever comes first.
Immune Duration Of Response (iDOR) | up to 4.5 years
  The time from first documentation of objective response to the first documentation of immune PD per immune RECIST or to death due to any cause, whichever comes first.
Progression Free Survival (PFS) evaluated by investigators | up to 4.5 years
  The time from start of study treatment to first documentation of objective PD per RECIST1.1 following study therapy, or to death due to any cause, whichever comes first.
Immune Progression Free Survival (iPFS) evaluated by investigators | up to 4.5 years
  The time from start of study treatment to first documentation of objective immune PD per immune RECIST following study therapy, or to death due to any cause, whichever comes first.
Overall Survival (OS) | up to 4.5 years
  The time from start of study treatment to date of death due to any cause.
Maximum serum concentration (Cmax) pharmacokinetics (PK) of ALE.C04 | up to 4.5 years
  Maximum serum concentration (Cmax) will be derived by non-compartmental analysis and summarized by dose cohort
Minimum serum concentration (Cmin) pharmacokinetics (PK) of ALE.C04 | up to 4.5 years
  Minimum serum concentration will be derived by non-compartmental analysis and summarized by dose cohort
Area under the concentration-time curve (AUC) pharmacokinetics (PK) of ALE.C04 | up to 4.5 years
  Area under the concentration-time curve will be derived by non-compartmental analysis and summarized by dose cohort
Maximum serum concentration (Cmax) Pharmacokinetics (PK) of pembrolizumab | up to 4.5 years
  Maximun Serum concentration (Cmax) by time point will be reported
Minimum serum concentration (Cmin) Pharmacokinetics (PK) of pembrolizumab | up to 4.5 years
  Minimum serum concentration (Cmin) by time point will be reported
Area under the concentration-time curve (AUC) Pharmacokinetics (PK) of pembrolizumab | up to 4.5 years
  Area under the concentration-time curve (AUC) by time point will be reported
Immunogenicity of ALE.C04 | up to 4.5 years
  To assess the presence of serum anti-drug antibodies (ADA) against ALE.C04
Change from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 | Phase II combination part only - Up to 4.5 year
  The C30 has 30 items in total. Among those items, 28 items are symptoms scales with score range from 1 to 4. A high score represents a high level of symptomatology. The 2 other items are global health status with score range of 1 to 7. A high score represents high quality of life.
Change from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Question Head and Neck module 43 (HN43) | Phase II combination part only - Up to 4.5 year
  The HN43 has 43 items of symptoms scale with score range of 1 to 4. A high score represents a high level of symptomatology.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Southern California USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Yale University Yale Cancer Center, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, Lake Saint Louis, Missouri
  - Gabrail Cancer Center Research, Canton, Ohio
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (3):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Hospitalier Saint-Andre, Bordeaux
  - Oncopole Claudius Regaud, Iuct-Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Prince Of Wales Hospital, Hong Kong, Hong Kong
- Italy (3):
  - Candiolo cancer Center,FPO IRCCS, Candiolo, Piedmont
  - Fondazione Irccs Istituto Nazionale Dei Tumori Di Milano, Milan
  - Istituto Europeo Di Oncologia S.R.L., Milan
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- Spain (4):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Incliva Biomedical Research Institute - Hospital Clinico Universitario Valencia, Valencia
- Inselspital, University Hospital Bern, Bern, Switzerland